CLINICAL TRIAL: NCT00590343
Title: An Open-label Phase II Study Evaluating the Safety and Efficacy of PTK787/ZK222584 in Patients With Metastatic Neuroendocrine Tumors That Have Evidence of Progressive Disease or an Increase in Disease Related Syndrome Symptoms.
Brief Title: Safety and Efficacy Study of PTK787/ZK222584 to Treat Metastatic Neuroendocrine Tumors
Acronym: PTK787
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Novartis (Industry)
Responsible Party: Lowell Anthony, MD, Louisiana State University Health Sciences Center-New Orleans
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTK787/ZK222584; LSU IRB-6355; NCT00627198 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Intervention=Patients will receive treatment with PTK787/ZK222584 daily. A treatment cycle will be defined as a 28-day period. Subjects will continue on their present treatment regimen of receiving Sandostatin LAR 30mg IM every 4 weeks.
  Interventions: Drug: vatalanib

INTERVENTIONS:
Drug: vatalanib — Subjects who meet all inclusion and exclusion criteria will receive an initial dose of PTK787/ZK222584 1,250mg once daily, and subjects will remain on the scheduled doses of Sandostatin LAR 30mg every 4 weeks.

SUMMARY:
The purpose of this study is to examine if PTK787/ZK222584 (vatalanib) will stabilize or decrease rising biochemical markers along with progressive disease or syndrome symptoms in patients with metastatic neuroendocrine tumors.

DETAILED DESCRIPTION:
This is an open-label, phase II study evaluating the safety and efficacy of PTK787/ZK222584 administered daily in subjects with neuroendocrine tumors that are experiencing progressive disease and/or whose tumor-related syndrome symptoms (flushing and diarrhea) are considered inadequately controlled despite optimal doses of octreotide therapy. Inadequate control is defined as a minimum of 2 flushing episodes or 6 bowel movements per day for 7 consecutive days. Subjects who meet all inclusion and exclusion criteria and have completed all baseline and screening testing will receive an initial dose of PTK787/ZK222584 1,250 mg once daily and subjects will also remain on the scheduled doses of Sandostatin LAR 30 mg every 4 weeks. Both drugs will be dosed on a flat schedule of mg, not by weight or body surface area. The PTK787/ZK222584 medication will be taken orally with daily dosing. Each tablet of PTK787/ZK 222584 is 250 mg. The subject will take five tablets of study medication per day 2 tabs am and 3 tabs pm. Subjects may continue to receive therapy as long as they do not experience unacceptable toxicities or evidence of disease progression as defined by RECIST criteria. Subjects will be evaluated with a daily log to assess the degree of symptom control (flushing and diarrhea) and subjects will be monitored every 2 weeks for 3 months then monthly for biochemical control and every three months for tumor response. Subjects will be monitored by the Investigator every two weeks for 3 months then monthly for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven metastatic neuroendocrine tumors (which extent is disease is determined by CT scan or MRI) and biochemical evidence of disease.
* Evidence of progressive disease or inadequate controlled disease related syndrome symptoms.
* Must be receiving Sandostatin LAR 30mg every 4 weeks
* Age >or= to 18 years old
* Karnofsky Performance Status > or = 60
* Measurable lesion(s) as per the modified RECIST criteria
* Laboratory values <or= 2 weeks prior to randomization: ANC >or= 1.5 x 10(9)/L, Platelets >or= 100 x 10 (9), Hemoglobin >or= 9g/dL, Serum creatinine <or= 1.5 ULN, Serum bilirubin <or= 1.5 ULN, Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) <or= 3.0 x ULN (<or= 5 x ULN if liver metastases present), Negative for proteinuria based on dip stick reading OR documentation of 1+ result for protein on dip stick reading, then total urinary protein <or= 500mg and measured creatinine clearance >or= 50ml/min from a 24 hour urine collection.
* Life expectancy >or= 12 weeks.
* Written informed consent obtained according to local guidelines.

Exclusion Criteria:

* Had previous radiolabeled somatostatin analog therapy within the last 6 months.
* Hepatic artery embolization within the last 6 months (1 month if there are other sites of measurable disease)
* Undergone cryoablation of hepatic metastasis within the last 2 months.
* History or presence of central nervous system (CNS) disease (ie:primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis)
* History of another primary malignancy <or= 5 years, with the exception of inactive basal or squamous cell carcinoma of the skin.
* Prior chemotherapy <or= 3 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities.
* Prior biologic or immunotherapy <or= 2 weeks prior to registration and/or randomization. Patients must have recovered from all therapy-related toxicities.
* Prior full field radiotherapy <or= 4 weeks or limited field radiotherapy <or= 2 weeks prior to randomization. Patients must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
* Major surgery (ie:laparotomy) <or= 4 weeks prior to randomization. Minor surgery <or= 2 weeks prior to randomization. Insertion of a vascular access device is not considered major or minor surgery in this regard. Patients must have recovered from all surgery-related toxicities.
* Patients who have received investigational drugs <or= 4 weeks prior to registration.
* Prior therapy with anti-VEGF agents
* Pleural effusion or ascites that causes respiratory compromise (>or= CTC grade 2 dyspnea)
* Female patients who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial in both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, therefore not considered effective for this study. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of study treatment.
* Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen.
* Unstable angina pectoris
* Symptomatic congestive heart failure
* Myocardial infarction <or= 6 months prior to registration
* Active or uncontrolled infection
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Chronic renal disease
* Subjects at risk of significant cardiac arrythmias
* Uncontrolled diabetes
* Acute or chronic liver disease (eg:hepatitis, cirrhosis)
* Impairment of gastrointestinal function or GI disease that may significantly alter absorption (ie:ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets.)
* Confirmed diagnosis of human immunodeficiency syndrome (HIV) infection are excluded at the investigator's discretion.
* Patients taking therapeutic warfarin sodium (Coumadin) or similar oral anticoagulants that are metabolized by the cytochrome P450 system. Heparin is allowed.
* Patients unwilling or unable to comply with the protocol.
* Known symptomatic gallstones
* Received glucocorticoid therapy within the past 6 months, or who are currently receiving any chemotherapeutic agents, insulin sensitizers (eg:metformin, pioglitazone, rosiglitazone), or exogenous growth hormones.
* Subjects with unacceptable concomitant diagnoses, or who have received medication and/or therapies (ie:illness or therapies that would place patient at increased risk, or would, in the opinion of the investigator, interfere with the evaluation of efficacy or safety.)
* Exhibit symptoms indicative of intolerance of Sandostatin LAR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-11; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in biochemical markers. | Quarterly= every 3 months

SECONDARY OUTCOMES:
Tumor response per triphasic CT scan. | Quarterly= every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lowell B Anthony, MD, Principal Investigator — Lousiana State University Health Sciences Center-NO
Locations (1):
- Neuroendocrine Clinic, Kenner, Louisiana, United States

REFERENCES:
- [Background] Drevs J, Muller-Driver R, Wittig C, Fuxius S, Esser N, Hugenschmidt H, Konerding MA, Allegrini PR, Wood J, Hennig J, Unger C, Marme D. PTK787/ZK 222584, a specific vascular endothelial growth factor-receptor tyrosine kinase inhibitor, affects the anatomy of the tumor vascular bed and the functional vascular properties as detected by dynamic enhanced magnetic resonance imaging. Cancer Res. 2002 Jul 15;62(14):4015-22. PMID 12124335